CLINICAL TRIAL: NCT02834728
Title: Frail Elderly Subjects: Inhospital Pathways and Adverse Outcome After Hospitalisation Via Emergency Department
Brief Title: Frail Elderly Subjects - Evaluation and Follow-Up
Acronym: SAFES Cohort
Status: Completed | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: 44N98
Record Dates: First submitted 2016-07-13; First posted 2016-07-15 (Estimated); Last update posted 2016-07-25 (Estimated); Status verified 2016-07

CONDITIONS: Frail Elderly People
MeSH Terms: interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Frail elderly people: A group of elderly people hospitalised in medical wards via emergency department
  Interventions: Behavioral: telephone interview

INTERVENTIONS:
Behavioral: telephone interview

SUMMARY:
This was a prospective multicenter cohort study of elderly people admitted to medical wards via emergency departments. Subjects were followed up to 36 months. It aimed to study the inhospital pathways and adverse geriatric outcomes. In all, 1306 subjects were included : 85+/-5 years, and mainly women (65%).

DETAILED DESCRIPTION:
The SAFES cohort was formed within a National Research Program (funded by the French Ministry of health) into the recruitment of emergency units in nine teaching hospitals. All nine centres had a geriatric ward. The inclusion of subjects ran from March 1st 2001 to January 17th 2002. To be eligible, patients were to be 75 or over, to have been hospitalised in a medical ward in the same hospital as the emergency unit to which they were initially admitted. Subjects were not eligible if hospitalisation was into intensive care or surgery, or if admission did not occur after admission to the emergency unit. Every day in each centre, patients admitted to the emergency unit were registered. From the list thus obtained, patients were selected by random draw stratified at two levels: in each week, 5 days were selected randomly, and for each of these days, two patients were chosen randomly. Next, each patient was visited by a specialist in geriatrics familiar with the survey procedures. In the course of this interview, patients were informed about the study, prior to signing the consent form. If the clinical status and/or the cognitive status of the patient did not enable informed consent, the interviewer referred to the subject's representative. Follow-up was by telephone interview after the 1st, 8th and 21st month and by face-to-face interviews after the 5th, 12th, 18th, and 24th month following the initial hospitalisation. Several outcome have been studied.

ELIGIBILITY:
Inclusion Criteria:

* Age of 75 years or over
* Admitted to medical ward via emergency department
* Consent to participate

Exclusion Criteria:

* Not hospitalised after emergency department stay
* Admitted to surgery or intensive car unit
* Died before signing informed consent form

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients were selected randomly from the emergency department. Subjects were to 75 years or over, and admitted to a medical ward after emargency department stay. Those who were admitted to surgery or intensive care units were excluded from the study
Sampling Method: Probability Sample
Enrollment: 1306 (Actual)
Dates: Start 2001-03; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Mortality | up to 36 months

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, France, Reims, France

REFERENCES:
- [Result] Tardieu E, Mahmoudi R, Novella JL, Oubaya N, Blanchard F, Jolly D, Drame M. [External validation of the short emergency geriatric assessment (SEGA) instrument on the SAFES cohort]. Geriatr Psychol Neuropsychiatr Vieil. 2016 Mar;14(1):49-55. doi: 10.1684/pnv.2016.0592. French. PMID 27005336
- [Result] de Boissieu P, Mahmoudi R, Hentzien M, Toquet S, Novella JL, Blanchard F, Jolly D, Drame M. Predictors of Long-Term Mortality in Oldest Old Patients (90+) Hospitalized to Medical Wards via the Emergency Department: The SAFES Cohort. J Nutr Health Aging. 2015 Jun;19(6):702-7. doi: 10.1007/s12603-015-0515-y. PMID 26054508
- [Result] Lang PO, Mahmoudi R, Novella JL, Tardieu E, Bertholon LA, Nazeyrollas P, Blanchard F, Jolly D, Drame M. Is obesity a marker of robustness in vulnerable hospitalized aged populations? Prospective, multicenter cohort study of 1 306 acutely ill patients. J Nutr Health Aging. 2014 Jan;18(1):66-74. doi: 10.1007/s12603-013-0352-9. PMID 24402392
- [Result] Narbey D, Jolly D, Mahmoudi R, Trenque T, Blanchard F, Novella JL, Drame M. Relationship between anticholinergic drug use and one-year outcome among elderly people hospitalised in medical wards via emergency department: the SAFES cohort study. J Nutr Health Aging. 2013 Sep;17(9):766-71. doi: 10.1007/s12603-013-0349-4. PMID 24154649
- [Result] Drame M, Lang PO, Novella JL, Narbey D, Mahmoudi R, Laniece I, Somme D, Gauvain JB, Heitz D, Voisin T, de Wazieres B, Gonthier R, Ankri J, Saint-Jean O, Jeandel C, Couturier P, Blanchard F, Jolly D. Six-month outcome of elderly people hospitalized via the emergency department: the SAFES cohort. Rev Epidemiol Sante Publique. 2012 Jun;60(3):189-96. doi: 10.1016/j.respe.2011.11.004. Epub 2012 May 16. PMID 22608011
- [Result] Dhaussy G, Drame M, Jolly D, Mahmoudi R, Barbe C, Kanagaratnam L, Nazeyrollas P, Blanchard F, Novella JL; SAFES Group. Is health-related quality of life an independent prognostic factor for 12-month mortality and nursing home placement among elderly patients hospitalized via the emergency department? J Am Med Dir Assoc. 2012 Jun;13(5):453-8. doi: 10.1016/j.jamda.2011.10.002. Epub 2011 Nov 13. PMID 22079488
- [Result] Drame M, Novella JL, Jolly D, Laniece I, Somme D, Heitz D, Gauvain JB, Voisin T, De Wazieres B, Gonthier R, Jeandel C, Couturier P, Saint-Jean O, Ankri J, Blanchard F, Lang PO. Rapid cognitive decline, one-year institutional admission and one-year mortality: analysis of the ability to predict and inter-tool agreement of four validated clinical frailty indexes in the SAFEs cohort. J Nutr Health Aging. 2011 Aug;15(8):699-705. doi: 10.1007/s12603-011-0164-8. PMID 21968868
- [Result] Lang PO, Drame M, Mahmoudi R, Jolly D, Laniece I, Saint-Jean O, Somme D, Heitz D, Gauvain JB, Voisin T, de Wazieres B, Gonthier R, Jeandel C, Couturier P, Ankri J, Blanchard F, Novella JL. [Frailty: learnings from the SAFEs cohort study and future perspectives for the research]. Geriatr Psychol Neuropsychiatr Vieil. 2011 Jun;9(2):135-49. doi: 10.1684/pnv.2011.0279. French. PMID 21690021
- [Result] Drame M, Fierobe F, Lang PO, Jolly D, Boyer F, Mahmoudi R, Somme D, Laniece I, Heitz D, Gauvain JB, Voisin T, De Wazieres B, Gonthier R, Ankri J, Saint-Jean O, Couturier P, Jeandel C, Blanchard F, Novella JL. Predictors of institution admission in the year following acute hospitalisation of elderly people. J Nutr Health Aging. 2011 May;15(5):399-403. doi: 10.1007/s12603-011-0004-x. PMID 21528168
- [Result] Drame M, Lang PO, Jolly D, Narbey D, Mahmoudi R, Laniece I, Somme D, Gauvain JB, Heitz D, Voisin T, de Wazieres B, Gonthier R, Ankri J, Saint-Jean O, Jeandel C, Couturier P, Blanchard F, Novella JL. Nursing home admission in elderly subjects with dementia: predictive factors and future challenges. J Am Med Dir Assoc. 2012 Jan;13(1):83.e17-20. doi: 10.1016/j.jamda.2011.03.002. Epub 2011 Apr 13. PMID 21493163
- [Result] Lang PO, Drame M, Jolly D, Novella JL, Blanchard F, Michel JP. [What do we learn from the SAFEs cohort to fit hospital care models for aged inpatient?]. Presse Med. 2010 Nov;39(11):1132-42. doi: 10.1016/j.lpm.2010.05.009. Epub 2010 Jul 1. French. PMID 20594791
- [Result] Somme D, Lazarovici C, Drame M, Blanc P, Lang PO, Gauvain JB, Voisin T, Gonthier R, De Wazieres B, Jeandel C, Couturier P, Blanchard F, Saint-Jean O. The geriatric patient: use of acute geriatrics units in the emergency care of elderly patients in France. Arch Gerontol Geriatr. 2011 Jan-Feb;52(1):40-5. doi: 10.1016/j.archger.2010.01.018. Epub 2010 Mar 3. PMID 20202700
- [Result] Lang PO, Zekry D, Michel JP, Drame M, Novella JL, Jolly D, Blanchard F. Early markers of prolonged hospital stay in demented inpatients: a multicentre and prospective study. J Nutr Health Aging. 2010 Feb;14(2):141-7. doi: 10.1007/s12603-009-0182-y. PMID 20126963
- [Result] Drame M, Dia PA, Jolly D, Lang PO, Mahmoudi R, Schwebel G, Kack M, Debart A, Courtaigne B, Laniece I, Blanchard F, Novella JL. [Factors predictive of long-term mortality in patients aged 75 years or older hospitalized from the emergency department: the SAFES cohort]. Presse Med. 2009 Jul-Aug;38(7-8):1068-75. doi: 10.1016/j.lpm.2009.01.019. Epub 2009 Apr 18. French. PMID 19376682
- [Result] Viatonou S, Drame M, Jolly D, Morrone I, Lang PO, Voisin T, Boyer FC, Schwebel G, Somme D, Blanchard F, Novella JL. Predictors of rapid cognitive decline among demented subjects aged 75 or more: ('Sujet Age Fragile--Evaluation et Suivi' Cohort-SAFES). Int J Geriatr Psychiatry. 2009 Jul;24(7):709-15. doi: 10.1002/gps.2183. PMID 19145574
- [Result] Prudent M, Drame M, Jolly D, Trenque T, Parjoie R, Mahmoudi R, Lang PO, Somme D, Boyer F, Laniece I, Gauvain JB, Blanchard F, Novella JL. Potentially inappropriate use of psychotropic medications in hospitalized elderly patients in France: cross-sectional analysis of the prospective, multicentre SAFEs cohort. Drugs Aging. 2008;25(11):933-46. doi: 10.2165/0002512-200825110-00004. PMID 18947261
- [Result] Drame M, Novella JL, Lang PO, Somme D, Jovenin N, Laniece I, Couturier P, Heitz D, Gauvain JB, Voisin T, De Wazieres B, Gonthier R, Ankri J, Jeandel C, Saint-Jean O, Blanchard F, Jolly D. Derivation and validation of a mortality-risk index from a cohort of frail elderly patients hospitalised in medical wards via emergencies: the SAFES study. Eur J Epidemiol. 2008;23(12):783-91. doi: 10.1007/s10654-008-9290-y. Epub 2008 Oct 21. PMID 18941907
- [Result] Drame M, Jovenin N, Novella JL, Lang PO, Somme D, Laniece I, Voisin T, Blanc P, Couturier P, Gauvain JB, Blanchard F, Jolly D. Predicting early mortality among elderly patients hospitalised in medical wards via emergency department: the SAFES cohort study. J Nutr Health Aging. 2008 Oct;12(8):599-604. doi: 10.1007/BF02983207. PMID 18810299
- [Result] Laniece I, Couturier P, Drame M, Gavazzi G, Lehman S, Jolly D, Voisin T, Lang PO, Jovenin N, Gauvain JB, Novella JL, Saint-Jean O, Blanchard F. Incidence and main factors associated with early unplanned hospital readmission among French medical inpatients aged 75 and over admitted through emergency units. Age Ageing. 2008 Jul;37(4):416-22. doi: 10.1093/ageing/afn093. Epub 2008 May 16. PMID 18487268
- [Result] Lang PO, Meyer N, Heitz D, Drame M, Jovenin N, Ankri J, Somme D, Novella JL, Gauvain JB, Couturier P, Laniece I, Voisin T, de Wazieres B, Gonthier R, Jeandel C, Jolly D, Saint-Jean O, Blanchard F. Loss of independence in Katz's ADL ability in connection with an acute hospitalization: early clinical markers in French older people. Eur J Epidemiol. 2007;22(9):621-30. doi: 10.1007/s10654-007-9150-1. Epub 2007 Jul 25. PMID 17653605
- [Result] Lang PO, Heitz D, Meyer N, Drame M, Jovenin N, Ankri J, Somme D, Novella JL, Gauvain JB, Colvez A, Couturier P, Laniece I, Voisin T, de Wazieres B, Gonthier R, Jeandel C, Jolly D, Saint-Jean O, Blanchard F. [Early indicators of prolonged hospitalization of the elderly: pilot study at Strasbourg University Hospital]. Presse Med. 2007 Mar;36(3 Pt 1):389-98. doi: 10.1016/j.lpm.2006.12.020. Epub 2007 Jan 17. French. PMID 17321360
- [Result] Lang PO, Heitz D, Hedelin G, Drame M, Jovenin N, Ankri J, Somme D, Novella JL, Gauvain JB, Couturier P, Voisin T, De Waziere B, Gonthier R, Jeandel C, Jolly D, Saint-Jean O, Blanchard F. Early markers of prolonged hospital stays in older people: a prospective, multicenter study of 908 inpatients in French acute hospitals. J Am Geriatr Soc. 2006 Jul;54(7):1031-9. doi: 10.1111/j.1532-5415.2006.00767.x. PMID 16866672